CLINICAL TRIAL: NCT03465722
Title: An International, Multicenter, Open-label, Randomized, Phase 3 Study of BLU-285 vs Regorafenib in Patients With Locally Advanced Unresectable or Metastatic Gastrointestinal Stromal Tumor (GIST)
Brief Title: (VOYAGER) Study of Avapritinib vs Regorafenib in Patients With Locally Advanced Unresectable or Metastatic GIST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Blueprint Medicines Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BLU-285-1303
Expanded Access: NCT03862885 (Approved for marketing)
Record Dates: First submitted 2018-03-07; First posted 2018-03-14 (Actual); Results first posted 2021-05-14 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-09

CONDITIONS: GIST
Keywords: Other Relapsed or Refractory Solid Tumors; BLU-285; BLU 285; BLUE-285; BLUE 285; Avapritinib; GIST imatinib relapse; GIST gleevec relapse; GIST KIT; GIST relapse; GIST refractory; GIST imatinib intolerance; GIST TKI treatment; GIST tyrosine kinase inhibitor treatment; GIST TKI; GIST tyrosine kinase inhibitor; Advanced GIST; GIST mutations; GIST treatments; Blueprint GIST; Relapsed GIST clinical trial; Refractory GIST clinical trial; KIT-mutant GIST; cancer gist; gastrointestinal stromal tumor; gist cancer; PDGFRA
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — avapritinib; regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- avapritinib (Experimental): 300 mg PO QD
  Interventions: Drug: avapritinib
- regorafenib (Active Comparator): 160 mg PO QD
  Interventions: Drug: regorafenib

INTERVENTIONS:
Drug: avapritinib — Avapritinib tablets for oral administration. Avapritinib will be dosed at 300 mg once daily, continuously.
  Other Names: BLU-285
  Arms: avapritinib
Drug: regorafenib — Regorafenib tablets for oral administration. Regorafenib will be dosed at 160 mg once daily for 3 weeks out of every 4 weeks (ie. 3 weeks on/1 week off).
  Other Names: Stivarga
  Arms: regorafenib

SUMMARY:
This is an open-label, randomized, Phase 3 study in patients with locally advanced unresectable or metastatic GIST (advanced GIST) of avapritinib (also known as BLU-285) versus regorafenib in patients previously treated with imatinib and 1 or 2 other TKIs.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are ≥ 18 years of age.
2. Patients who have histologically confirmed metastatic or unresectable GIST.
3. Patients who received imatinib and 1 or 2 other TKIs as prior treatment regimens. Patients who experienced intolerance to prior therapies must have objective disease progression prior to enrollment onto BLU-285-1303 study.
4. Patients who have an Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 to 1.

Exclusion Criteria:

1. Patients who have received prior treatment with avapritinib or regorafenib.
2. Patients who have previously received more than 3 different TKI treatment regimens.
3. Patients who are known to be both V-kit Hardy-Zuckerman 4 feline sarcoma viral oncogene homolog (KIT) and platelet-derived growth factor receptor alpha (PDGRFα) wild type.
4. Patients who received any systemic anticancer therapy within 1 week before the first dose of study drug.
5. Patients who have clinically significant cardiovascular disease
6. Patients have experienced arterial thrombotic or embolic events within 6 months before the first dose of study drug, or venous thrombotic events within 14 days of the first dose of study drug
7. Patients who have experienced any hemorrhage or bleeding event NCI CTCAE version 5.0 Grade 3 or higher within 4 weeks before the first dose of study drug
8. Patients who have a known risk of intracranial bleeding, or a history of intracranial bleeding within 1 year prior to the first dose of study drug
9. Patients who have a symptomatic non-healing wound, ulcer, gastrointestinal perforation, or bone fracture.
10. Patients who have poor organ function as defined by laboratory parameters specified in the protocol.
11. Patients who have received neutrophil growth factor support within 14 days of first dose of study drug.
12. Patients who require therapy with a concomitant medication that is a strong inhibitor or strong inducer of CYP3A4.
13. Patients who have had a major surgical procedure within 14 days of the first dose of study drug. Patient has significant traumatic injury within 28 days before the first dose of study drug.
14. Patients who have a history of another primary malignancy that has been diagnosed or required therapy within 3 years before first dose of study drug.
15. Patients who have a history of a seizure disorder requiring anti-seizure medication.
16. Patients who have metastases to the brain.
17. Patients who have a QT interval corrected using Fridericia's formula (QTcF) of > 450 msec.
18. Women who are unwilling, if not postmenopausal or surgically sterile, to abstain from sexual intercourse or employ highly effective contraception from the time of the first dose of study drug and for at least 60 days after the last dose of study drug. Men who are unwilling, if not surgically sterile, to abstain from sexual intercourse or employ highly effective contraception from the time of the first dose of study drug and for at least 90 days after the last dose of study drug.
19. Women who are pregnant.
20. Women who are breastfeeding.
21. Patients who have prior or ongoing clinically significant illness, medical condition, surgical history, physical finding, or laboratory abnormality as determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 476 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2021-09-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (114):
- United States (30):
  - Mayo Clinic Cancer Center, Phoenix, Arizona
  - UCLA Hematology/Oncology - Santa Monica, Santa Monica, California
  - University of Colorado Hospital, Aurora, Colorado
  - Rocky Mountain Cancer Centers, Boulder, Colorado
  - Washington Hospital Center - Oncology and Hematology, Washington D.C., District of Columbia
  - Mayo Clinic Cancer Center, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Northside Hospital, Atlanta, Georgia
  - Northwestern Medicine, Chicago, Illinois
  - The University of Chicago Medical Center, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Washington University in Saint Louis, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - OHSU - Knight Cancer Institute, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Tennessee Oncology, Nashville, Tennessee
  - USO - Texas Oncology, Dallas, Texas
  - Texas Oncology - Denton South, Denton, Texas
  - University of Texas MD Anderson, Houston, Texas
  - Texas Oncology - Waco, Waco, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Summit Cancer Centers, Spokane, Washington
  - Medical College of Wisconsin - Froedtert Hospital, Milwaukee, Wisconsin
- Australia (3):
  - Flinders Medical Center, Adelaide
  - Monash Health, Clayton
  - The Canberra Hospital, Garran
- AKH, Klinik f. Innere Med. I, Onkologie, Vienna, Austria
- Belgium (2):
  - Institut Jules Bordet, Brussels
  - Leuven Cancer Institute, Leuven
- Canada (3):
  - Cross Cancer Institute, Edmonton, Alberta
  - University Health Network, Toronto, Ontario
  - Jewish General Hospital, Montreal
- China (19):
  - Beijing Cancer Hospital, Beijing
  - Chinese PLA General Hospital, Beijing
  - West China Hospital Sichuan University, Chengdu
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - Fujian Medical University Union Hospital, Fuzhou
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou
  - The Sixth Affiliated Hospital of Sun Yat-Sen University, Guangzhou
  - The First Affiliated Hospital, Zhejiang University, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - The First Affiliated Hospital of Nanchang Medical University, Nanchang
  - Guangxi Medical University Affiliated Tumor Hospital & Oncology Medical College, Nanning
  - The Affiliated Hospital of Qingdao University, Qingdao
  - Fudan University Shanghai Cancer Center, Shanghai
  - Fudan University Zhongshan Hospital, Shanghai
  - Shanghai Jiaotong University School of Medicine, Renji Hospital, Shanghai
  - Liaoning Cancer Hospital & Institute, Shenyang
  - Tianjin Cancer Hospital, Tianjin
  - Affiliated Cancer Hospital of Xinjiang Medical University, Ürümqi
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
- Czechia (2):
  - Onkologická klinika Fakultní nemocnice Olomouc, Olomouc
  - Fackultni Nemocnice v Motole, Prague
- France (8):
  - Institut Bergonié, Bordeaux
  - Centre Oscar Lambret, Lille
  - UNICANCER - Lyon, Centre Léon-Bérard, Lyon
  - Institute Paoli Calmettes, Marseille
  - La Timone University Hospital, Marseille
  - Institut Curie, Paris
  - Centre Rene Gauducheau, Saint-Herblain
  - Gustave Roussy Cancer Campus, Villejuif
- Germany (7):
  - HELIOS Klinikum Bad Saarow, Bad Saarow
  - HELIOS Klinikum Berlin-Buch, Berlin
  - Medizinische Fakultät Carl Gustav Carus, Dresden
  - Universitaetsklindum Essen, Essen
  - Universitätsklinikum Frankfurt, Frankfurt
  - Studienzentrale GbR Lübecker Onkologische Schwerpunktpraxis Dres. med. Uthgenannt, Lübeck
  - Rupercht-Karls-Universitaet Heidelberg, Mannheim
- Hungary (4):
  - Fovarosi Onkormanyzat Szent Laszlo Korhaz, Budapest
  - Magyar Honvédség Egészségügyi Központ Onkológiai Osztály, Budapest
  - Medical Oncology University Debrecen, Debrecen
  - University of Pécs, Pécs
- Italy (7):
  - Azienda Ospedaliero Universitaria Sant'Orsola Malpighi, Bologna
  - Candiolo Cancer Institute - FPO, IRCCS, Candiolo
  - AOUC Azienda Ospedaliero - Universitaria Careggi, Florence
  - Fondazione IRCCS Istituto Nazionale dei Tumori Milano, Milan
  - Istituto Europeo di Oncologia, Milan
  - Universita degli Studi di Palermo - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone, Palermo
  - Campus Bio-Medico - Oncology Medica, Roma
- Netherlands (3):
  - Nederlands Kanker Instituut - Antoni Van Leeuwenhoek Ziekenhuis, Amsterdam
  - Radboud University Medical Center, Nijmegen
  - Erasmus Medical Center, Rotterdam
- Poland (4):
  - Sanodzielny Publiczny Zaklad Opieki Zdrowotnej Szpital Uniwesytecki w Krakowie, Oddzial Kliniczny Onkologii, Krakow
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej MSWiA z W-MCO, Olsztyn
  - Maria Skodowska Curie Memorial Cancer Centre and Institute of Oncology, Warsaw
  - Dolnoslaskie Centrum Onkologii we Wrocawiu, Wroclaw
- National Cancer Centre Singapore, Singapore, Singapore
- South Korea (5):
  - Ajou University Hospital, Suwon, Gyeong Gi-do
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
- Spain (9):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Institut Català d'Oncologia - Hospital Duran i Reynals, Barcelona
  - Vall d'Hebron, Barcelona
  - Hospital La Paz, Madrid
  - Hospital Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Virgen del Rocio, Seville
  - Fundacion Instituto Valenciano de Oncologia, Servicio de Oncologia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Skanes University Hospital, Lund, Sweden
- United Kingdom (5):
  - Beatson West of Scotland Cancer Centre, Glasgow
  - The Royal Marsden Hospital, London
  - Guy's Hospital, London
  - The Christie NHS Foundation Trust, Manchester
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield

REFERENCES:
- [Derived] Serrano C, Bauer S, Gomez-Peregrina D, Kang YK, Jones RL, Rutkowski P, Mir O, Heinrich MC, Tap WD, Newberry K, Grassian A, Shi H, Bialick S, Schoffski P, Pantaleo MA, von Mehren M, Trent JC, George S. Circulating tumor DNA analysis of the phase III VOYAGER trial: KIT mutational landscape and outcomes in patients with advanced gastrointestinal stromal tumor treated with avapritinib or regorafenib. Ann Oncol. 2023 Jul;34(7):615-625. doi: 10.1016/j.annonc.2023.04.006. Epub 2023 Apr 25. PMID 37105265
- [Derived] Kang YK, George S, Jones RL, Rutkowski P, Shen L, Mir O, Patel S, Zhou Y, von Mehren M, Hohenberger P, Villalobos V, Brahmi M, Tap WD, Trent J, Pantaleo MA, Schoffski P, He K, Hew P, Newberry K, Roche M, Heinrich MC, Bauer S. Avapritinib Versus Regorafenib in Locally Advanced Unresectable or Metastatic GI Stromal Tumor: A Randomized, Open-Label Phase III Study. J Clin Oncol. 2021 Oct 1;39(28):3128-3139. doi: 10.1200/JCO.21.00217. Epub 2021 Aug 3. PMID 34343033
- [Derived] Gebreyohannes YK, Wozniak A, Zhai ME, Wellens J, Cornillie J, Vanleeuw U, Evans E, Gardino AK, Lengauer C, Debiec-Rychter M, Sciot R, Schoffski P. Robust Activity of Avapritinib, Potent and Highly Selective Inhibitor of Mutated KIT, in Patient-derived Xenograft Models of Gastrointestinal Stromal Tumors. Clin Cancer Res. 2019 Jan 15;25(2):609-618. doi: 10.1158/1078-0432.CCR-18-1858. Epub 2018 Oct 1. PMID 30274985

RESULTS

PARTICIPANT FLOW:
Groups:
- Avapritinib: 300 mg PO QD avapritinib: Avapritinib tablets for oral administration. Avapritinib will be dosed at 300 mg once daily, continuously.
- Regorafinib: 160 mg PO QD regorafenib: Regorafenib tablets for oral administration. Regorafenib will be dosed at 160 mg once daily for 3 weeks out of every 4 weeks (ie. 3 weeks on/1 week off).
Period: Overall Study
Arm/Group | Avapritinib | Regorafinib
Started | 240 | 236
Completed | 0 | 0
Not Completed | 240 | 236
Not completed — Withdrawal by Subject | 21 | 14
Not completed — Death | 89 | 87
Not completed — Lost to Follow-up | 5 | 3
Not completed — Administrative/Other | 33 | 32
Not completed — Not treated | 1 | 2
Not completed — Sponsor decision | 91 | 98

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Avapritinib | Regorafinib | Total
Number analyzed (Participants) | 240 | 236 | 476
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (10.96) | 61.0 (10.74) | 61.1 (10.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 80 | 158
  Male | 162 | 156 | 318
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 64 | 64 | 128
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 9 | 5 | 14
  White | 139 | 143 | 282
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 27 | 23 | 50
Region of Enrollment [Number; unit: participants]
  Singapore | 2 | 2 | 4
  Hungary | 2 | 1 | 3
  United States | 71 | 62 | 133
  Czechia | 3 | 1 | 4
  United Kingdom | 12 | 12 | 24
  Spain | 14 | 11 | 25
  Canada | 2 | 6 | 8
  Austria | 0 | 1 | 1
  Netherlands | 2 | 6 | 8
  South Korea | 23 | 20 | 43
  Sweden | 6 | 7 | 13
  Belgium | 1 | 1 | 2
  China | 35 | 39 | 74
  Poland | 10 | 9 | 19
  Italy | 13 | 15 | 28
  Australia | 5 | 5 | 10
  France | 22 | 20 | 42
  Germany | 17 | 18 | 35
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per meter square] — Both height and weight measurements are needed for body mass index calculation. Some patients had missing height and/or weight measurements. Only patients with both a height and a weight measurement are included in the body mass index calculation Population: Both height and weight measurements are needed for body mass index calculation. Some patients had missing height and/or weight measurements. Only patients with both a height and a weight measurement are included in the body mass index calculation
  kilogram per meter square
    number analyzed (Participants) | 230 | 225 | 455
    (all) | 25.50 (5.563) | 24.69 (5.163) | 25.10 (5.378)

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Avapritinib Based on Progression-free Survival (PFS) Determined by Central Radiological Assessment Per Modified Response Evaluation Criteria in Solid Tumors (mRECIST), Version 1.1
Description: To demonstrate the efficacy of avapritinib based on progression-free survival (PFS) determined by central radiological assessment per modified Response Evaluation Criteria in Solid Tumors (mRECIST), version 1.1 in patients with advanced GIST following 2 or 3 regimens of prior treatment with a tyrosine kinase inhibitor (TKI), including imatinib, compared to patients treated with regorafenib. A progressively growing tumor must meet the following criteria: a) the target lesions must be greater or equal to 2cm in size and be a new GIST active lesion or b) the target lesions must be expanding on at least 2 sequential imaging studies.
Time Frame: 24 Months
Population: Intent-to-Treat Population that included all patients randomized to study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avapritinib | Regorafinib
Number analyzed (Participants) | 240 | 236
months | 4.2 [3.7 to 5.6] | 5.6 [3.8 to 7.2]

2. Secondary Outcome: Objective Response Rate (ORR) Determined by Central Radiology Assessment Per mRECIST, Version 1.1
Description: To evaluate objective response rate (ORR) determined by central radiology assessment per mRECIST, version 1.1 in patients with advanced GIST treated with avapritinib compared to patients treated with regorafenib. A complete response (CR) per modified Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) is defined as complete disappearance of all target lesions. A partial response (PR) is defined as at least 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum of diameters. Overall Response (OR) = CR + PR
Time Frame: 24 Months
Population: Intent-to-Treat Population that included all patients randomized to study.
Measure: Count of Participants; unit: Participants
Arm/Group | Avapritinib | Regorafinib
Number analyzed (Participants) | 240 | 236
Participants
  Responder | 41 | 17
  Non-Responder | 199 | 219

3. Secondary Outcome: Overall Survival (OS) in Patients With Advanced GIST Treated With Avapritinib Compared to Patients Treated With Regorafenib
Description: To evaluate overall survival (OS) in patients with advanced GIST treated with avapritinib compared to patients treated with regorafenib
Time Frame: 24 Months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avapritinib | Regorafinib
Number analyzed (Participants) | 240 | 236
months | 19.2 [19.2 to NA] — Since the primary endpoint of statistically significant improvement in PFS was not met patients are not being followed for OS. The upper bound of the confidence interval is not estimable by the Kaplan-Meier analysis due to the short follow-up time. | 17.4 [15.8 to NA] — Since the primary endpoint of statistically significant improvement in PFS was not met patients are not being followed for OS. The upper bound of the confidence interval is not estimable by the Kaplan-Meier analysis due to the short follow-up time.

4. Secondary Outcome: European Organisation for Research and Treatment of Cancer Quality of Life (EORTC-QLQ-30). Change in Individual Scores in Patients With Advanced GIST Treated With Avapritinib Compared to Patients Treated With Regorafenib
Description: The Global Health Status Score is derived from question 29 and 30 on the EORTC-QLQ-C30 tool. The change in score was assessed between baseline and week 12 in patients treated with advanced GIST treated with avapritinib compared to patients treated with regorafenib. The Global Health Status Score score range is 0 to 100 with a higher score indicating better global health status. A positive change indicates improvement in global health status.
Time Frame: Difference between baseline and week 12 of treatment
Population: Intent-to-Treat Population with both a baseline and a Week 12 measurements.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Avapritinib | Regorafinib
Number analyzed (Participants) | 123 | 138
scores on a scale | -5.7 (24.29) | -4.4 (20.74)

ADVERSE EVENTS:
Time Frame: From the date of first study drug administration to 30 days after last study drug administration, approximately 6 months
Description: The total number of at risk patients includes patients that were randomized to treatment and received at least one dose of treatment. Patients that were randomized by did not receive treatment were excluded from the safety analysis.
Arm/Group | Avapritinib | Regorafinib
All-Cause Mortality (participants affected / at risk) | 89/239 | 87/234
Serious Adverse Events (participants affected / at risk) | 106/239 | 91/234
Other Adverse Events (participants affected / at risk) | 218/239 | 224/234
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Avapritinib (N=239) | Regorafinib (N=234)
Anaemia (Blood and lymphatic system disorders) | 27 | 7
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 0
Myocarditis (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 0 | 1
Retinal vein occlusion (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 13 | 11
Ascites (Gastrointestinal disorders) | 5 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 6 | 5
Vomiting (Gastrointestinal disorders) | 5 | 2
Diarrhoea (Gastrointestinal disorders) | 4 | 5
Gastric haemorrhage (Gastrointestinal disorders) | 4 | 1
Abdominal distension (Gastrointestinal disorders) | 2 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 3
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Diverticular perforation (Gastrointestinal disorders) | 1 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 2
Gastrointestinal fistula (Gastrointestinal disorders) | 2 | 0
Intestinal obstruction (Gastrointestinal disorders) | 2 | 3
Intestinal perforation (Gastrointestinal disorders) | 2 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 | 1
Inguinal hernia strangulated (Gastrointestinal disorders) | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Small intestine ulcer (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 0 | 1
Disease progression (General disorders) | 3 | 1
Face oedema (General disorders) | 2 | 0
Generalised oedema (General disorders) | 2 | 0
Multi-organ failure (General disorders) | 3 | 1
Pyrexia (General disorders) | 4 | 7
Chest pain (General disorders) | 1 | 1
Fatigue (General disorders) | 2 | 2
General physical health deterioration (General disorders) | 3 | 0
Hernia perforation (General disorders) | 1 | 0
Hyperthermia (General disorders) | 1 | 0
Inflammation (General disorders) | 1 | 0
Asthenia (General disorders) | 0 | 3
Condition aggravated (General disorders) | 1 | 1
Malaise (General disorders) | 0 | 2
Non-cardiac chest pain (General disorders) | 0 | 1
Hepatic haemorrhage (Hepatobiliary disorders) | 3 | 0
Jaundice (Hepatobiliary disorders) | 2 | 0
Portal hypertension (Hepatobiliary disorders) | 2 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hepatic pain (Hepatobiliary disorders) | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Sepsis (Infections and infestations) | 5 | 0
Bacteraemia (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 2 | 2
Lung infection (Infections and infestations) | 1 | 1
Peritonitis (Infections and infestations) | 1 | 0
Rhinovirus infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 3
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Anastomotic stenosis (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Amylase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 1
Neutrophil count decreased (Investigations) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 2
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Liver carcinoma ruptured (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour fistulisation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Cognitive disorder (Nervous system disorders) | 3 | 1
Haemorrhage intracranial (Nervous system disorders) | 2 | 0
Transient ischaemic attack (Nervous system disorders) | 2 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Coma (Nervous system disorders) | 1 | 1
Facial paresis (Nervous system disorders) | 0 | 1
VIIth nerve paralysis (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 1
Major depression (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 4 | 4
Autoimmune nephritis (Renal and urinary disorders) | 1 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash morbilliform (Skin and subcutaneous tissue disorders) | 0 | 1
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 3
Gastric mucosal lesion (Gastrointestinal disorders) | 0 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Peritoneal sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Enteritis infectious (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Avapritinib (N=239) | Regorafinib (N=234)
Periorbital oedema (Eye disorders) | 68 | 0
Lacrimation increased (Eye disorders) | 45 | 0
Eyelid oedema (Eye disorders) | 35 | 0
Dyspepsia (Gastrointestinal disorders) | 21 | 16
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 16 | 7
Dry mouth (Gastrointestinal disorders) | 7 | 15
Stomatitis (Gastrointestinal disorders) | 7 | 40
Oedema peripheral (General disorders) | 55 | 13
Mucosal inflammation (General disorders) | 3 | 28
Conjunctivitis (Infections and infestations) | 12 | 0
White blood cell count decreased (Investigations) | 42 | 7
Aspartate aminotransferase increased (Investigations) | 33 | 33
Weight decreased (Investigations) | 24 | 53
Blood creatinine increased (Investigations) | 21 | 12
Weight increased (Investigations) | 18 | 4
Alanine aminotransferase increased (Investigations) | 15 | 29
Blood alkaline phosphatase increased (Investigations) | 6 | 13
Hypocalcaemia (Metabolism and nutrition disorders) | 15 | 11
Hypoalbuminaemia (Metabolism and nutrition disorders) | 12 | 16
Hypomagnesaemia (Metabolism and nutrition disorders) | 11 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 16
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 | 25
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 22
Dizziness (Nervous system disorders) | 32 | 19
Memory impairment (Nervous system disorders) | 31 | 5
Headache (Nervous system disorders) | 29 | 43
Dysgeusia (Nervous system disorders) | 20 | 11
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 8 | 71
Hair colour changes (Skin and subcutaneous tissue disorders) | 33 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 24 | 38
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 15
Dry skin (Skin and subcutaneous tissue disorders) | 10 | 18
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 | 14
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 4 | 143
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 13
Anxiety (Psychiatric disorders) | 12 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-06-20): https://cdn.clinicaltrials.gov/large-docs/22/NCT03465722/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-01): https://cdn.clinicaltrials.gov/large-docs/22/NCT03465722/SAP_001.pdf